CLINICAL TRIAL: NCT01128114
Title: A 4-week, Multi-Centre, Open-label, Non-comparative, Phase IV Study of the Broad Clinical Benefit for Seroquel XR (Quetiapine Fumarate Extended Release) With Flexible Dose as an add-on Therapy in the Treatment of Acute Bipolar Mania Patients With Partial Response to Current Therapy
Brief Title: Study of the Broad Clinical Benefit for Seroquel XR With Flexible Dose as an add-on Therapy in the Treatment of Acute Bipolar Mania Patients With Partial Response to Current Therapy
Acronym: RELEASE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00080
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Results first posted 2012-04-10 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Acute Bipolar Mania
Keywords: Acute bipolar mania; Seroquel XR; Quetiapine fumarate; Add-on therapy
MeSH Terms: interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quetiapine XR (Experimental): Quetiapine fumarate (Seroquel XR)
  Interventions: Drug: Quetiapine fumarate (Seroquel XR)

INTERVENTIONS:
Drug: Quetiapine fumarate (Seroquel XR) — Extended Release(XR) 50 mg, 200 mg, 300 mg and/or 400 mg tablet, oral, once daily in the evening, from assignment to the end of the study.
  Other Names: Seroquel XR tablet

SUMMARY:
The primary objective of this study is to evaluate the broad clinical benefit of dosing Seroquel XR with flexible in the treatment of acute bipolar mania patients with partial response to existing therapy. Clinical benefit will be assessed with the Clinical Global Impression-Clinical Benefit (CGI-CB) score, according to a classification based on the principles outlined in the CGI efficacy index. Improvement in clinical benefit will be defined as a decrease from baseline in CGI-CB.

DETAILED DESCRIPTION:
A 4-week, Multi-Centre, Open-label, Non-comparative, Phase IV Study of the Broad Clinical Benefit for Seroquel XR (Quetiapine Fumarate Extended Release) With Flexible Dose as an add-on Therapy in the Treatment of Acute Bipolar Mania Patients With Partial Response to Current Therapy

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical diagnosis meeting the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria (1. Bipolar I Disorder, manic or mixed type with/without psychotic feature, 2. Diagnosis should be confirmed by the Mini Inte)
* Currently on Lithium/Valproate without antipsychotics more than 3 weeks consecutive treatment YMRS total score ≥16 at study entry

Exclusion Criteria:

* Non-response to antipsychotic treatments for manic symptoms in previous episodes
* A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria (1. Unstable DM defined as enrolment glycosylated hemoglobin (HbA1c) >8.5%, 2. Admitted to hospital for treatment of DM or DM related illness in past 12 weeks, etc)
* An absolute neutrophil count (ANC) of 1.5 x 10^9 per liter

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joon Woo Bahn, Study Chair — AstraZeneca; Won-Myong Bahk, MD, Principal Investigator — St.Mary's hospital, The Catholic University of Korea
Locations (11):
- South Korea (11):
  - Research Site, Junam, Choongnam
  - Research Site, Cheonan, Chungcheongnam-do
  - Research Site, Chuncheon, Gangwondo
  - Research Site, Bucheon-si, Gueonggido
  - Research Site, Suwon, Gyeonggi-do
  - Research Site, Gyeongju, Gyeongsangbuk-do
  - Research Site, Yongsan-gu, Seoul
  - Research Site, Daejeon
  - Research Site, Gyungbook
  - Research Site, Naju
  - Research Site, Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- Quetiapine XR: Extended Release (XR) 50mg, 200mg 300mg and/or 400mg tablet, oral once daily in the evening, from assignment to the end of the study
Period: Overall Study
Arm/Group | Quetiapine XR
Started | 32
Completed | 24
Not Completed | 8
Not completed — Treatment Withdrawn | 6
Not completed — Screening Failed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Quetiapine XR
Number analyzed (Participants) | 32
Age, Customized [Number; unit: participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 0
  Unknown | 5
Sex/Gender, Customized [Number; unit: participants]
  Unknown | 4
  Male | 10
  Female | 18
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 32

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients With Improvement From Baseline to Week 4 in Clinical Global Impression-Clinical Benefit Score (LOCF)
Description: CGI-CB is used to evaluate the investigator's global weighted impression of efficacy and interference of adverse event from baseline to every visit. Improvement in clinical benefit is defined as a decrease from baseline in CGI-CB. Rank 1 denotes best possible benefit from new treatment and rank 10 indicates that there is no benefit from treatment.
Time Frame: Baseline, week 4
Population: As the study was terminated prematurely none of the randomized patients have been analysed.
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR
Number analyzed (Participants) | 0

2. Secondary Outcome: The Mean Change From Baseline to Week 4 in - YMRS (Young Mania Rating Scale) Total Score
Description: The YMRS is an 11-item, multiple-choice diagnostic questionnaire which psychiatrists use to measure severity of manic episodes. There are 4 items graded on a 0 to 8 scale (irritability, speech, thought content, disruptive/aggressive behavior), and 7 items graded on 0 to 4 scale. These 4 items are given twice the weight of the others to compensate for poor cooperation from severely ill patients. Typical YMRS baseline scores can vary a lot. They depend on patients' clinical features such as mania (YMRS = 12), depression (YMRS = 3), or euthymia (YMRS = 2.
Time Frame: Baseline, week 4
Reporting Status: Not Posted

3. Secondary Outcome: The CGI-I (Clinical Global Impression-Improvement of Illness) Change From Baseline to Week 4
Description: The Global Improvement scale (CGI-I) is scored to rate the patient's change from baseline CGI. A CGI-I score of 1 indicates that a patient is "very much improved" and a score of 7 indicates that a patient is "very much worse." CGI-I scores greater than 4 indicate worsening, while scores less than 4 indicate improvement. At all following visits CGI-I will also be rated. The following calculations will be made: Proportion of patients with CGI Global Improvement rating ≤ 2 at Day 29
Time Frame: Baseline, week 4
Reporting Status: Not Posted

4. Secondary Outcome: The Mean Change From Baseline to Week 4 in CGI-S (Clinical Global Impression-Severity of Illness) Score
Description: The CGI-S is scored to rate patient's current clinical state. At enrolment patient's condition is rated using the CGI-S. At assignment CGI-S is again completed and a score of at least 4 (moderately ill). The score at assignment Day 1 will be regarded as the baseline value. At all following visits CGI-S will be rated. Each CGI item is scored on a scale from 1 to 7. A CGI-S score of 1 indicates that a patient is "Normal, not at all ill" and a score of 7 indicates that a patient is "Among the most extremely ill patients".
Time Frame: Baseline, week 4
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Quetiapine XR
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

LIMITATIONS AND CAVEATS:
In March 2011, considering the low patient inclusion rate (32 patients recruited so far whereas study objective was 125 patients for 85 completers), the study was ended prematurely earlier than the planned date. No analysis was conducted afterwards.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No